CLINICAL TRIAL: NCT05469009
Title: Assessment of Safety and Feasibility of Exablate Blood-Brain Barrier Disruption for the Treatment of Patients With With Mild Cognitive Impairment (MCI) or Mild Alzheimer's Disease (AD) Undergoing Standard of Care Monoclonal Antibody (mAb) Therapy
Brief Title: Safety and Feasibility of Exablate Blood-Brain Barrier Disruption for Mild Cognitive Impairment or Mild Alzheimer's Disease Undergoing Standard of Care Monoclonal Antibody (mAb) Therapy
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ali Rezai (Other)
Collaborators: InSightec (Industry)
Responsible Party: Sponsor-Investigator, Ali Rezai, Neurosurgeon, West Virginia University
Organization: West Virginia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2110449196
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease 1
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer disease type 1 | interventions — aducanumab; lecanemab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Infusion plus Exablate BBBO Treatment (Experimental): Intravenous infusion of Aducanumab or Lecanemab every 2-4 weeks (per standard of care) followed by blood brain barrier opening by FUS.
  Interventions: Drug: Aducanumab; Device: Exablate Model 4000 Type 2; Drug: Lecanemab

INTERVENTIONS:
Drug: Aducanumab — Standard aducanumab therapy will be given by intravenous infusion every 4 weeks for 6 cycles with blood brain barrier opening
  Other Names: Aduhelm
Device: Exablate Model 4000 Type 2 — The Exablate Model 4000 will be utilized for the BBBO (blood-brain barrier opening) after each cycle of Aducanumab or Lecanemab administered per label.
  Other Names: Focused Ultrasound
Drug: Lecanemab — Standard lecanemab therapy will be given by intravenous infusion every 2 weeks for up to 6 cycles with blood brain barrier opening
  Other Names: Leqembi

SUMMARY:
The purpose of this study is to assess the safety and feasibility of administering standard of care monoclonal antibody (mAb) infusion therapy in combination with opening the blood-brain barrier with the Exablate Model 4000 Type 2 device in patients with mild Alzheimer's disease (AD) or mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
The primary objectives of this study is to evaluate the safety and feasibility of BBBO (blood-brain barrier opening) using the Exablate Model 4000 Type 2 in the setting of standard aducanumab or lecanemab therapy among patients with mild cognitive impairment (MCI) or mild Alzheimer's disease (AD) with confirmed β-amyloid, who are eligible for aducanumab or lecanemab infusion therapy, and to also evaluate the safety of the BBO procedure through patient examination (neurological and cognitive/behavioral) and MRI assessments during the treatment and follow-up.

The secondary objectives of this study is to determine the effect of BBBO in patients with MCI or mild AD treated with aducanumab or lecanemab on brain β-amyloid plaque measured by amyloid positron emission tomography (PET), as well as to assess the clinical impact of BBBO with standard aducanumab or lecanemab therapy, if any, as assessed with ADAS Cog 11 and MMSE over time following BBBO.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give informed consent
* Probable mild cognitive impairment due to AD
* Modified Hachinski Ischemia Scale (MHIS) score of <= 4
* Mini Mental State Exam (MMSE) scores > 21+.
* Short form Geriatric Depression Scale (GDS) score of <= 7
* Amyloid PET scan consistent with the presence of β-amyloid (A+)
* Able to communicate sensations during the Exablate MRgFUS procedure
* Able to attend all study visits (i.e., life expectancy of 1 year or more)

Exclusion Criteria:

* MRI findings:
* Significant cardiac disease or unstable hemodynamic status
* History of a liver disease, bleeding disorder, coagulopathy or a history of spontaneous hemorrhage
* Known cerebral or systemic vasculopathy
* Significant depression (GDS > 7) and/or at potential risk of suicide (C-SSRS > 2)
* A severity score of 2 or more on any of the 'Delusions', 'Hallucinations' or 'Agitation/Aggression' subscales of the Neuropsychiatry Inventory (NPI-Q)
* Known sensitivity/allergy to gadolinium(gadobutrol), DEFINITY or its components, or 18F-florbetaben.
* Known hypersensitivity to DEFINITY or its components.
* Any contraindications to MRI scanning
* Untreated, uncontrolled sleep apnea
* History of untreated or uncontrolled seizure disorder or epilepsy.
* Impaired renal function
* Does not have a reliable caregiver
* Currently in a clinical trial involving an investigational product or non-approved use of a drug or device or in any other type of medical research.
* Respiratory: chronic pulmonary disorders
* History of clinically significant recent drug or alcohol use disorder who may be at higher risk for seizure or infection.
* Positive human immunodeficiency virus (HIV) which can lead to increased entry of HIV into the brain parenchyma leading to HIV encephalitis.
* Potential blood-borne infections, which can lead to increased entry to brain parenchyma leading to meningitis or brain abscess.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Treatment intervention related adverse events | From baseline, up to 5 year post last treatment
  The total number of adverse events following each treatment through end of the study
Treatment intervention related serious adverse events | From baseline, up to 5 year post last treatment
  The total number of serious adverse events following each treatment through end of the study

SECONDARY OUTCOMES:
Beta-Amyloid plaques within the brain | From baseline, up to 5 year post last treatment
  Beta-Amyloid uptake value measured by Amyloid PET scan
Cognitive performance (ADAS COG 11) | From baseline, up to 5 year post last treatment
  Change in cognitive performance using the Alzheimer's Disease Assessment Cognitive Subscale, rating scores from 0-70. The greater the dysfunction, the greater the score. A score of 70 represents the most severe impairment and 0 represents the least impairment.
Cognitive performance (MMSE) | From baseline, up to 5 year post last treatment
  Change in cognitive performance using the Mini Mental Status Exam, rating scores from 0-30. 25 or higher being classed as normal. A score below 24 is considered abnormal, indicating possible cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rezai, MD, FAANS, Principal Investigator — WVU Rockerfeller Neuroscience Institute
Locations (1):
- West Virginia University Rockefeller Neuroscience Institute, Morgantown, West Virginia, United States